CLINICAL TRIAL: NCT03501745
Title: Through Remote Management and Propaganda of Intelligent Mobile Phone, the Standard Rate of Blood Pressure Control and the Change of Renal Function Were Observed
Brief Title: Smart-CKD/BP Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Qinghai University (Other)
Responsible Party: Principal Investigator, Pengli Luo, Deputy chief physician, Affiliated Hospital of Qinghai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20180330
Record Dates: First submitted 2018-03-30; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-03

CONDITIONS: CKD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Management Group (Other)
  Interventions: Behavioral: WeChat
- control group (Other)
  Interventions: Behavioral: WeChat

INTERVENTIONS:
Behavioral: WeChat — Through remote management and propaganda of intelligent mobile phone, the standard rate of blood pressure control and the change of renal function were observed.

SUMMARY:
Through remote management and propaganda of intelligent mobile phone, the standard rate of blood pressure control and the change of renal function were observed.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis in line with the 2012 international kidney disease: improving global outcomes (kidney disease improving global out-comes, KDIGO) of chronic kidney disease diagnosis standard of hypertension diagnosis, "China Hypertension Prevention Guide 2010" diagnostic criteria;
2. and will have the use of intelligent mobile phone, and a network connection;
3. at the age of 18-70.

Exclusion Criteria:

1. GFR<15 ml/min or start replacement therapy;
2. do not understand Chinese, do not understand Chinese;
3. malignant tumor patients;
4. have mental illness;
5. there is consciousness disorder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Control rate of blood pressure control | 1 year
  Average blood pressure of each patient ,thenStatistics of the number of blood pressure control standards .
Drug compliance | 1 year
  Take medications according to the doctor's advice

CONTACTS AND LOCATIONS:
Locations (1):
- Pengli Luo, Qinghai, Xining, China

IPD SHARING:
Plan to Share IPD: Undecided